CLINICAL TRIAL: NCT05828706
Title: The Effects of Pain and Disability Resulting From Shoulder Pathologies On Balance and Mobility
Status: Completed | Type: Observational
Sponsor: Biruni University (Other)
Collaborators: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Guzin Kaya Aytutuldu, PhD, Biruni University
Other Study IDs: Biruni Univ
Record Dates: First submitted 2023-04-12; First posted 2023-04-25 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2023-06

CONDITIONS: Shoulder Injuries
Keywords: balance; shoulder pain; mobility; functionality
MeSH Terms: conditions — Shoulder Injuries; Shoulder Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Among the musculoskeletal pathologies, shoulder pain is the most common symptom after back and neck pain (1, 2). One out of every three adults experiences shoulder pain and limitation in shoulder movements, which affects the functionality of the patients and leads to disability. (2) Impairment of one or more sensory inputs coming from the visual, somatosensory or afferent pathways from the vestibular system (3-4) causes deterioration of balance control and falls (4-5). Since pain affects the somatosensory system, it causes a decrease in balance ability. This study will be conducted to examine the effect of pain and functionality on balance in shoulder pathologies. Our study included pathologies such as impingement, rotator cuff syndrome, frozen shoulder, fracture between November 1, 2022 and January 1, 2023; A total of 40 patients, 18 females and 12 males, between the ages of 41-74 (56.30±9.25) will be included. Sociodemographic information form, Shoulder Pain and Disability Index (SPADI), One-leg standing test, 5 sit and stand test, TINetti balance and walking test will be evaluated for the included patients. SPSS Version 21.0 program was used for statistical analysis. With Pearson Correlation analysis, it will be evaluated whether the data are related or not.

DETAILED DESCRIPTION:
Upper extremity pathologies are musculoskeletal problems that are common in the community, resulting in loss of work force and negative continuation of recreational activities (1,2). Among the pathologies of the musculoskeletal system, shoulder pain is the most common symptom after back and neck pain (3, 4). One out of every three adults experiences shoulder pain and limitation in shoulder movements, which affects the functionality of the patients and leads to disability (4). Among these common problems, there are many diseases such as rotator cuff injuries, adhesive capsulitis, acromioclavicular joint degenerations, calcific tendinitis and instability (5). Impairment of one or more sensory inputs coming from the visual, somatosensory or afferent pathways from the vestibular system (6-7) causes deterioration of balance control and falls (7-8). Since pain affects the somatosensory system, it causes a decrease in balance ability. In addition, pain-induced balance control and muscle inhibition pathways share some pathways in the central nervous system (9 ,10). Therefore, muscle inhibition mechanisms caused by pain may negatively affect balance ability (10,11). It has been proven that patients with shoulder pain have deficiencies in shoulder proprioception as well as trunk and lower extremity coordination (10,12). Problem-free and painless upper extremity movements are mostly related to the stability of the trunk and this is closely related to the stability of the lower extremities and balance control. Any deficiency in trunk and lower extremity stability is largely tolerated by compensating the structures around the upper extremity by increasing speed and power, and this situation paves the way for upper extremity pathologies. It remains unclear whether the lack of balance is a cause or a consequence of injury in individuals with shoulder problems (13). Myers et al. reported that proprioception and coordination deficiencies greatly affect shoulder problems, therefore somatosensory deficiencies in the lower extremity and trunk may cause problems in the upper extremity region (14). Other known factors affecting balance, apart from proprioception and coordination, are attention (15,16), age (17,18), gender and body mass index (BMI) (19,20). Decreased balance can lead to limitation of movement, falls and injuries (21). This situation may also require rehabilitation of balance problems caused by upper extremity pathologies. There is very little published research investigating the relationship between different levels of shoulder pain, balance ability, risk of falling, and fear of falling, covering all age groups diagnosed with musculoskeletal shoulder problems. Although it has been shown that the balance of patients with shoulder pain is adversely affected, it is not clear how pain level and disability affect balance parameters. Therefore, in this study, it was aimed to investigate the relationship between pain severity, functionality and balance in shoulder pathologies,

ELIGIBILITY:
Inclusion Criteria:

1. Having a pathology related to the upper extremity shoulder such as Impingement, Rotator cuff tear or repair, Adhesive capsulitis (frozen shoulder),
2. Able to communicate
3. Individuals between the ages of 40-65 who agreed to participate in the study

Exclusion Criteria:

1. Having vision and hearing problems
2. Having other accompanying neurological, psychiatric and/or orthopedic problems other than shoulder pathologies
3. Having a pregnancy status

Ages: 41 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Our study was carried out by Prof. Dr. Bezmialem Vakif University Faculty of Medicine, Department of Physical Medicine and Rehabilitation. Dr. It is planned to include patients referred by Teoman Aydın. In our study, post-hoc power analysis was performed and it was determined that 36 individuals were needed to achieve 95% power with an effect size of r:0.50. Considering the possibility of cases dropping out of the study, it is planned to include 40 individuals.
  Sociodemographic information form, Shoulder Pain and Disability Index (SPADI), One-leg standing test, 5 sit and stand test, TINetti balance and walking test will be evaluated for the included patients.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-05-26 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
Evaluation of Shoulder Pain and Functionality (SPADI) | 10 minutes
  SPADI includes 5 questions about pain and 8 questions about disability, and patients are asked to answer these questions on a numerical scale (22). The score is calculated for pain and disability separately and together. While calculating the score, the sum of the points given to the questions in each section is divided by the maximum score that can be obtained from that section and multiplied by 100. Similarly, in the total score, the total score of all questions is divided by 130 and multiplied by 100. Thus, the scores obtained as a percentage range from 0 to 100.
One Leg Stance Test | 10 minutes
  The one-leg stance test is a test that measures the time of standing on the right and left extremities of the patient and evaluates the static balance. Evaluation is made by recording the time from the moment the patient starts to stand on one leg to the first moment when postural stability is impaired (25). It gives an idea about an individual's risk of falling. If he can stand on one leg for 30 seconds, it can be said that the test is over. If the cut-off value is <10 seconds, it means "unbalance", and if it is <5 seconds, it means "there is a risk of falling" (26).
5 Repetition Sit and Stand Test | 10 minutes
  It is a performance test that evaluates the functional strength of the lower extremity, transitional movements, fall risk, and dynamic balance by recording the performance of individuals sitting and standing on a chair 5 times in series (27). Whitney et al. Developed by The patient is asked to quickly stand up and sit down from the standard chair in which he sits with his arms crossed over his shoulders and his back leaning against the chair (28). Norm times according to age are '60-69' 11.4 seconds, '70-79' 12.6 seconds, and '80-89' 14.8 seconds. The periods indicating the presence of risk of falling are 'Old >12 sec. (If >15 repetitive), Vestibular disease >15 sec., Parkinson's >16 sec' (29).

CONTACTS AND LOCATIONS:
Locations (1):
- Prof. Dr. Bezmialem Vakif University Faculty of Medicine, Department of Physical Medicine and Rehabilitation., Istanbul, Turkey (Türkiye)